CLINICAL TRIAL: NCT03129399
Title: Nasal Intubation Using the King Vision Video Laryngoscope:a Randomized,Controlled Comparison With McGrath MAC Video Laryngoscope
Brief Title: Comparison of King Vision Video Laryngoscope to McGrath MAC Video Laryngoscope for Nasal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Sun Yu, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: suny
Record Dates: First submitted 2017-04-14; First posted 2017-04-26 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Nasal Intubation
Keywords: anesthesia; King Vision; videolaryngoscope; nasotracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- King Vision video laryngoscope (Experimental)
  Interventions: Device: King Vision video laryngoscope
- McGrath MAC video laryngoscope (Active Comparator)
  Interventions: Device: McGrath MAC video laryngoscope

INTERVENTIONS:
Device: King Vision video laryngoscope — nasal intubation using King Vision video laryngoscope Device after general anesthesia induction
  Arms: King Vision video laryngoscope
Device: McGrath MAC video laryngoscope — nasal intubation with McGrath MAC video laryngoscope Device after general anesthesia induction
  Arms: McGrath MAC video laryngoscope

SUMMARY:
This study was designed to determine the comparison between the King Vision video laryngoscope and McGrath MAC video laryngoscope for nasotracheal intubation.Patients were divided into 2 groups of 40 patients each.Patients of King Vision group [n=40]and Macintosh group [n=40]were intubated using respective devices.This study is the first to search the use of King Vision video laryngoscope for nasotracheal intubation in difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Scheduled for general anesthesia with nasotracheal intubation
* Cormach-Lehane score 3-4

Exclusion Criteria:

* contraindications to nasal intubation
* Patients with a history of anti-hypertensive drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-05-20 (Estimated); Study Completion 2018-06-20 (Estimated)

PRIMARY OUTCOMES:
time to intubation | 0 min after nasal intubation
  from taking of the intubation device to successful intubation

SECONDARY OUTCOMES:
Hemodynamic changes | 1 min before general anesthesia induction
  heart rate
Hemodynamic changes | 1 min after general anesthesia induction
  heart rate
Hemodynamic changes | 3 min after general anesthesia induction
  heart rate
Hemodynamic changes | 5 min after general anesthesia induction
  heart rate
ease of intubation | 5 min after nasal intubation
  VAS scores
incidence of trauma | 24hour after surgery
  sore throat, hoarseness, etc
incidence of trauma | 1hour after surgery
  sore throat, hoarseness, etc
number of failures | 5 min after nasal intubation
  intubation failure
the degree of Cormach-Lehane | 5 min after nasal intubation
  glottic exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital,Affililated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China